# The Effects of Video-Assisted Breastfeeding Education Given to Primiparous Pregnant Women on Breastfeeding Self-Efficacy: Randomised Control Study

## **Study Protocol**

Before initiating the study, ethics committee approval (27.05.2022 dated and 2022-506 numbered decision) was obtained from the Ondokuz Mayıs University Social and Humanities Research Ethics Committee where the study was (see Appendix 1). Before the data collection form was applied, the purpose of the study was explained to all participants and written consent was obtained from those who volunteered to participate in the study. (see Appendix 2-3).

## Statistical Analysis Plan

Data were evaluated by using IBM SPSS v.23 (IBM Corp. Armonk, NY, USA) program and presented with descriptive statistics such as "number, percentage, arithmetic mean, standard deviation". Chi-square test for categorical variables and independent sample t-test for continuous variables were used to confirm the differences in demographic and obstetric characteristics between groups. Independent sample t-test was used for intergroup comparison of PBSES scores and paired sample t-test was used for intragroup comparison. Statistical significance value was accepted as p<0.05.

## **Appendix 1 Ethics Committee Approval**



#### ONDOKUZ MAYIS ÜNİVERSİTESİ SOSYAL VE BEŞERİ BİLİMLER ARAŞTIRMALARI ETİK KURUL KARARLARI

| KARAR TARİHİ | TOPLANTI SAYISI | KARAR SAYISI |
|--------------|-----------------|--------------|
| 27.05.2022 | 5 | 2022-506 |

KARAR NO: 2022-506 Üniversitemiz Sağlık Bilimleri Fakültesi Öğr. Gör. Ayşe METİN ile Dr. Öğr. Üyesi Nazlı BALTACI'nın "Primipar Gebelere Verilen Video Destekli Emzirme Eğitiminin Emzirme Öz Yeterliliğe Etkisi" isimli öğretim üyesi araştırmasına (bilimsel araştırma) ilişkin anket ve ölçek çalışmalarını içeren 63855 sayılı dilekçesi okunarak görüşüldü.

Üniversitemiz Sağlık Bilimleri Fakültesi Öğr. Gör. Ayşe METİN ile Dr. Öğr. Üyesi Nazlı BALTACI'nın "Primipar Gebelere Verilen Video Destekli Emzirme Eğitiminin Emzirme Öz Yeterliliğe Etkisi" isimli öğretim üyesi araştırmasına (bilimsel araştırma) ilişkin anket ve ölçek çalışmalarının kabulüne oy birliği ile karar verildi.

## **Appendix 2 Informed voluntary consent form (Experimental Group)**

Hello, my name is XXX. I am a lecturer at Ondokuz Mayıs University, Faculty of Health Sciences, and a doctoral student in the Department of Nursing. Ondokuz Mayıs University, Faculty of Health Sciences, Department of Nursing, I am conducting my research titled " The Effects of Video-Assisted Breastfeeding Education Given to Primiparous Pregnant Women on Breastfeeding Self-Efficacy: Randomised Control Study".

The aim of this study is to determine the effects of online video-assisted breastfeeding education on breastfeeding self-efficacy in primiparous pregnant women. Within the scope of the research, video-supported breastfeeding education in an online classroom (<a href="https://meet.google.com/zsd-ions-gsw">https://meet.google.com/zsd-ions-gsw</a>) for 6-8 people and individual counselling via phone and Whatsapp application. If you do not want to continue the research, you can leave at any time. Your data may be used for publication purposes without disclosing your name. Participation in the research is entirely voluntary. Reading and approving this form will mean that you agree to participate in the research.

Consent to Participate in the Study

I have read all the explanations in the Informed Volunteer Consent Form. Written and verbal explanations about the research whose subject and purpose are stated above were made to me by the researcher named below. I had the opportunity to ask questions and discuss and received satisfactory answers. I know that I can quit this study whenever I want, without having to give any reason, and that I will not face any negative consequences if I quit. I agree to participate in this research voluntarily, without any pressure or coercion.

History: Participant: Signature Researcher: XXX Signature:

## **Appendix 3 Informed voluntary consent form (Control Group)**

Hello, my name is XXX. I am a lecturer at Ondokuz Mayıs University, Faculty of Health Sciences, and also a doctoral student in the Department of Nursing. Ondokuz Mayıs University, Faculty of Health Sciences, Department of Nursing, Lecturer Prof. Dr. I am conducting my thesis research titled "The Effect of Nursing Counseling Based on Neuman Systems Model on Perceived Stress, Coping with Stress and Birth Outcomes in Pregnant Women at Risk of Preterm Labor" under the supervision of YYY.

This study aims to determine the effect of education and counseling offered to pregnant women at risk of premature birth on stress perception, coping with stress and pregnancy outcomes. In line with the results of this research, it is aimed to provide education and counseling to pregnant women at risk of premature birth. The research will be conducted through a survey of approximately 10-15 minutes. The surveys will be administered 3 times in total until birth. If you do not want to continue the research, you can leave at any time. Everything you say during the interview will remain confidential. Your name and personal information will be used solely for research purposes and will never be disclosed to others. Your data may be used for publication purposes without disclosing your name. Participation in the research is entirely voluntary. Reading and approving this form will mean that you agree to participate in the research.

## Consent to Participate in the Study

I have read all the explanations in the Informed Volunteer Consent Form. Written and verbal explanations about the research whose subject and purpose are stated above were made to me by the researcher named below. I had the opportunity to ask questions and discuss and received satisfactory answers. I know that I can quit this study whenever I want, without having to give any reason, and that I will not face any negative consequences if I quit. The research in question is carried out on its own, without any pressure or coercion.

| History: |
|--------------|
| Participant: |
| Signature |
| Researcher: |
| XXX |
| Signature: |